CLINICAL TRIAL: NCT04309266
Title: Understanding the Impact of Robot Assisted Therapy and Metacognitive Skills Training on Functional Performance for Children With Hemiparesis: A Pilot Study
Brief Title: The Impact of Robot Assisted Therapy and Metacognitive Skills Training for Children With Hemiparesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: MGH Institute of Health Professions (Other)
Responsible Party: Principal Investigator, Casey Rabideau, Primary Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB P00032628
Record Dates: First submitted 2020-03-04; First posted 2020-03-16 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Hemiparesis; Hemiplegic Cerebral Palsy; Hemiparesis;Poststroke/CVA
Keywords: arm weakness; cerebral palsy; stroke; in utero; cognition; occupational therapy; robot therapy; robot assisted therapy; metacognition; children; pediatric; Amadeo; arm; upper extremity; Tyromotion; ALPS; motor learning; rehabilitation
MeSH Terms: conditions — Paresis; Cerebral Palsy; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Robot Assisted Therapy with Metacognitive Skills Training (Experimental): All participants will be enrolled in the single arm of this study, where they will receive robot assisted therapy combined with metacognitive skills training.
  Interventions: Device: Amadeo by Tyromotion; Behavioral: Active Learning Protocol for Stroke

INTERVENTIONS:
Device: Amadeo by Tyromotion — Distal upper extremity/hand robot for robot-assisted therapy
Behavioral: Active Learning Protocol for Stroke — Metacognitive approach involving active problem solving for using the affected upper extremity in motoric activities. Also includes a home program.
  Other Names: ALPS

SUMMARY:
The Occupational Therapy Department at Boston Children's Hospital is teaming up with MGH Institute of Health Professions to explore the benefits of using robot assisted therapy (Amadeo) and a problem solving approach (Active Learning Program for Stroke) to achieving functional goals for children ages 7-17 years old that have hemiparesis. The hope is to help participants make gains in both hand/arm skills and progress in everyday activities such as self-care, play, school and work. Participation will look like regular therapy with sessions 3 times weekly for 8 weeks. Each visit will include time for games on the Amadeo and time spent problem solving current activity challenges for each child. Families are encouraged to participate.

DETAILED DESCRIPTION:
Robot assisted therapy and Active Learning Program for Stroke (ALPS) are unique interventions that are feasible and effective for individuals with neuromotor impairments. To the best of our knowledge, this is a novel intervention approach and thus there are no preliminary studies to acknowledge that reference this combined technique. There have been studies which evaluated the Amadeo and metacognitive approaches in isolation, but not combined.

The goal of this pilot study is to better understand the impact of a combined approach using both robot assisted therapy and metacognitive skills training through ALPS on the functional performance outcomes of children with hemiparesis. Our primary aim is to evaluate the feasibility of this pilot study intervention as measured by adequate recruitment of necessary population, participant attendance to scheduled sessions, participant adherence to home program and clinician competence/adherence with protocol administration. Our secondary aim is to understand the preliminary impact of a combined approach to intervention involving robot-assisted therapy and a metacognitive strategy training ALPS on upper limb motor skills and function of children with hemiparesis. It is hypothesized that utilizing this combined bottom-up and top-down approach will be a feasible option for intervention and that preliminary outcomes will be promising. If successful, this project has the potential to improve rehabilitation and habilitation outcomes of children with hemiparesis.

This study will be set as a prospective pilot study with pre- and post-intervention and one month follow-up evaluation. Study procedures will occur within Boston Children's Hospital's Department of Physical and Occupational Therapy Service. For the duration of this trial, participants will not be allowed to participate in additional occupational therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child must be between 7 and 17 years of age at the start of the study.
* Child must have hemiparesis with at least partial active grasp and release.
* Child must be able to follow multi-step commands.
* Child must have a caregiver available who can assist with implementation of home exercise program.
* Child must speak English.
* Child must have hemiparesis caused by cerebral vascular accident.
* Child must have adequate insurance to cover evaluation, re-evaluations, and intervention, as this study will be billed to participants' insurance.

Exclusion Criteria:

* Child must not have received botulinum toxin or phenol injections within 4 months of and/or during intervention.
* Child must have tone less than 3/4 on Modified Ashworth Scale.
* Child must not be considered legally blind.
* Child must not have contraindications for use of robot assisted device (ie. recent fracture or skin lesion).
* Child must not be non-verbal.
* Child must have not had reconstructive surgery to the affected upper extremity within the last year.
* Child must not be receiving active oncology plan of care.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Patient Recruitment | Determined at the conclusion of the study, approximately 2 years
  Quantitative tracking of patient recruitment - was the goal n of 15 children with hemiparesis who completed the study attained?
Implementation of Intervention | Determined at the conclusion of the study, approximately 2 years
  Was the recommended frequency/duration of Amadeo and ALPS provided to participants?
Implementation of Intervention | Determined at the conclusion of the study, approximately 2 years
  Did patients adhere to daily home programming? - At least 80% compliance will be deemed successful.
Staff's Perceived Competency of Hemiparesis | Determined at the conclusion of the study, approximately 2 years
  Measured by a post-training survey.
Staff's Actual Competency of Hemiparesis | Every 3 months until conclusion of the study, up to 2 years
  Measured by routine audits.
Staff's Perceived Competency of Amadeo | Determined at the conclusion of the study, approximately 2 years
  Measured by post-training survey.
Staff's Actual Competency of Amadeo | Every 3 months until conclusion of the study, up to 2 years
  Measured by routine audits.
Staff's Actual Competency of Amadeo | Determined at the conclusion of the study, approximately 2 years
  Measured by fidelity checklist.
Staff's Perceived Competency of ALPS | Determined at the conclusion of the study, approximately 2 years
  Measured by post-training survey.
Staff's Actual Competency of ALPS | Every 3 months until conclusion of the study, up to 2 years
  Measured by routine audits.
Staff's Actual Competency of ALPS | Determined at the conclusion of the study, approximately 2 years
  Measured by fidelity checklist.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * Administered to all participants. The parent/caregiver and child will collaboratively develop goal priority areas. Both the parent/caregiver and child will then separately score performance and satisfaction in each identified area so that both parent and child perception are obtained.
  * Provides data for participant's self-perceived performance capacity and satisfaction with performance on self-determined functional goal areas.
  * Performance and Satisfaction are ranked on a scale of 1-10, with higher scores signifying higher self-perceived performance/satisfaction in personally identified meaningful activities.
  * Parent/Child interview with performance/satisfaction score rankings completed
  * Administration time = ~15 minutes
Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT): Activities of Daily Living and Social/Cognitive Domains | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * Administered to all participants. To be completed by child's parent/caregiver.
  * Provides data for a participant's level of independence with Activities of Daily Living (ADLs)
  * Parent/Child questionnaire
  * Items in Activities of Daily Living and Social/Cognitive domains scored on scale of 1-4, with higher scores signifying increased ease in tasks.
  * Administration time = ~15 minutes, can be completed prior to clinic evaluation.
Box & Blocks | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * Administered to all participants
  * Provides data regarding a child's gross manual dexterity
  * Measures number of blocks transferred from one compartment to the next in 60 seconds.
  * Administration time = ~10 minutes
Jebsen Hand Function Test | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * Administered to all participants
  * Provides data regarding the uni-manual skills required for ADLs.
  * Scores are timed measurements
  * Administration time = ~15-30 minutes
9 Hole Peg Test | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * Administered to participants who are successful to pick up small manipulatives as part of Jebsen
  * Provides data regarding fine manual dexterity
  * Scores are timed measurements. Participants will be allowed maximum 4 minutes for trial with hemiparetic upper extremity.
  * Administration time = ~10 minutes

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Upper Extremity Full Version | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * Administered to all participants, completed by parent/guardian
  * Provides data for a participant's level of upper extremity function within a variety of functional tasks including ADLS, Instrumental Activities of Daily Living (IADLs), Education.
  * Parent/Child questionnaire
  * All items rated on scale of either 1-5 or 1-4, with higher scores signifying higher levels of independence.
  * Administration time = ~15 minutes
Quality of Upper Extremity Skills Test (QUEST) | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * All participants evaluated for subsections A (dissociated movements) and B (Grasps)
  * Provides data regarding dissociated movement and grasp patterns
  * No formal score acquired within this study. QUEST will be used as a way to have universal language for grasp and pinch between providers.
Shriner's Hospital Upper Extremity Evaluation (SHUEE) | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * Administered to all participants
  * Provides data regarding the spontaneous use of a hemiparetic upper extremity and the dynamic segmental alignment of the extremity while performing tasks on demand.
  * Scores are calculated in percentiles.
  * Spontaneous Functional Analysis items scored on scale of 0-5, with higher scores signifying more spontaneous use of the affected arm.
  * Dynamic Positional Analysis items ranked on scale of 0-3, with higher scores signifying optimal alignment of the respective arm segment (elbow, forearm, wrist, finger, thumb).
  * Grasp and Release Analysis items scored on scale of 0-3, with higher scores signifying optimal alignment of the wrist in grasp/release tasks.
  * Administration time = ~15 minutes
Pain Scale | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * All participants evaluated
  * Provides data on participant's current pain level.
  * Ranked using 0-10 numeric scale, with higher rankings signifying increased level of pain.
  * Administration time = ~1 minute
Stereognosis Sensory Testing | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * All participants evaluated
  * Measures child's ability to perceive and recognize an object in hand. Scored in percentile correct.
Two-Point Discrimination Sensory Testing | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * All participants evaluated
  * Two-Point Discrimination - ability to discern that two nearby objects touching the skin are truly two distinct points, not one. Score in percentile correct.
Active and Passive Range of Motion | Administered at week 1, week 10 of protocol (after completing 8 weeks of the intervention), and week 14 (1 month after week 10).
  * All participants evaluated for shoulder flexion, abduction, external rotation and internal rotation, elbow flexion/extension, forearm supination/pronation, wrist flexion/extension and gross grasp/release measurements.
  * Measured with goniometer in degrees
  * Administration time = ~15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Rabideau, MS, OTR, BCP, Principal Investigator — Department of Physical and Occupational Therapy Service
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data including patient age and performance on outcome measures will be shared with Susan Fasoli, ScD, OTR/L at MGH Institute of Health Professions via RedCap online database. Susan will assist with data analysis and write-up of findings.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Present (3/2020) - until study write-up is prepared for publishing (anticipated fall 2022).